CLINICAL TRIAL: NCT07116395
Title: Outcomes of Tranexamic Acid With Anticoagulants in Orthopaedic Trauma Procedures: A Prospective Study
Brief Title: Prospective Study: TXA, Anticoagulant, Orthopaedic Trauma
Acronym: TXA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Arbi Nazarian, MD (Other)
Collaborators: Inspire Health Medical Group (Unknown)
Responsible Party: Sponsor-Investigator, Arbi Nazarian, MD, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nazarian_TXA_Prospective2025
Record Dates: First submitted 2025-07-29; First posted 2025-08-11 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: Patients Undergoing Operative Fixation of Long Bone Fractures Within the Community Medical Centers System
Keywords: TXA; Anticoagulant; Orthopaedic Trauma
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Yes TXA Administered (Experimental)
  Interventions: Drug: Tranexamic Acid (TXA)
- No TXA Administered (No Intervention)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — orthopedic trauma patients who are on anticoagulation
  Arms: Yes TXA Administered

SUMMARY:
Tranexamic acid, an anti-fibrinolytic agent, is commonly given after induction of general anesthesia in patients undergoing hip and knee arthroplasty. This medication has been associated with decreased blood loss during these procedures, decreased rate of blood transfusion, decreased hospital costs, and no increased risk of thrombotic complication. Given the safety and efficacy of this medication in one subspeciality of orthopedics, it is warranted to investigate the use of it in another subspeciality where blood loss is also of concern. It is also of the utmost importance to identify medications that can safely be given to our population to not only improve patient outcomes but also decrease patient costs in the setting of significant disparities. The application of these findings to orthopedic trauma is not something that has been largely studied or appears in the literature. We hope to fill this gap of knowledge to allow for the application of a safe and beneficial medication to a much larger subset of patients than that that is already receiving the medication routinely. The use of TXA in orthopedic patients who are on anticoagulation versus those who are not is also not something that has been previously studied and another knowledge gap that we hope to fill.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing operative fixation of long bone fractures; Included conditions include femoral neck fractures, intertrochanteric femur fractures, femoral shaft fractures, distal femur fractures, and tibial shaft fractures that undergo surgical management

Exclusion Criteria:

* Exclusion criteria for this study will be patients under 18 and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimated blood loss (EBL) comparison between those who received TXA vs no TXA | EBL note is made post-procedure by surgical team, and research team will collect data at least one month post-procedure
  Less estimated blood loss after surgery for patients who were administered TXA

SECONDARY OUTCOMES:
Hospital Length of Stay for Patients who received TXA vs no TXA | EBL note is made post-procedure by surgical team, and research team will collect data at least one month post-procedure
  Patient medical records will be reviewed post-operatively and data will be collected in our study specific data sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Arbi Nazarian, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share IPD with other researchers as the study team does not have full approval to share data from our local collaborative hospital site.

REFERENCES:
- [Background] Lin YK, Liu KT, Chen CW, Lee WC, Lin CJ, Shi L, Tien YC. How to effectively obtain informed consent in trauma patients: a systematic review. BMC Med Ethics. 2019 Jan 23;20(1):8. doi: 10.1186/s12910-019-0347-0. PMID 30674301
- [Background] Ockerman A, Vanassche T, Garip M, Vandenbriele C, Engelen MM, Martens J, Politis C, Jacobs R, Verhamme P. Tranexamic acid for the prevention and treatment of bleeding in surgery, trauma and bleeding disorders: a narrative review. Thromb J. 2021 Aug 11;19(1):54. doi: 10.1186/s12959-021-00303-9. PMID 34380507
- [Background] Zhang P, Liang Y, Chen P, Fang Y, He J, Wang J. Combined application versus topical and intravenous application of tranexamic acid following primary total hip arthroplasty: a meta-analysis. BMC Musculoskelet Disord. 2017 Feb 21;18(1):90. doi: 10.1186/s12891-017-1429-0. PMID 28222709
- [Background] Zhu Q, Yu C, Chen X, Xu X, Chen Y, Liu C, Lin P. Efficacy and Safety of Tranexamic Acid for Blood Salvage in Intertrochanteric Fracture Surgery: A Meta-Analysis. Clin Appl Thromb Hemost. 2018 Nov;24(8):1189-1198. doi: 10.1177/1076029618783258. Epub 2018 Jun 21. PMID 29929380
- [Background] Deng ZF, Zhang ZJ, Sheng PY, Fu M, Xu DL, He AS, Liao WM, Kang Y. Effect of 3 different anticoagulants on hidden blood loss during total hip arthroplasty after tranexamic acid. Medicine (Baltimore). 2020 Sep 4;99(36):e22028. doi: 10.1097/MD.0000000000022028. PMID 32899057
- [Background] Hourlier H, Fennema P. Tranexamic acid use and risk of thrombosis in regular users ofantithrombotics undergoing primary total knee arthroplasty: a prospectivecohort study. Blood Transfus. 2018 Jan;16(1):44-52. doi: 10.2450/2016.0160-16. Epub 2016 Oct 4. PMID 27723454
- [Background] Hunt BJ. The current place of tranexamic acid in the management of bleeding. Anaesthesia. 2015 Jan;70 Suppl 1:50-3, e18. doi: 10.1111/anae.12910. PMID 25440395